CLINICAL TRIAL: NCT03425383
Title: Association of Endodontic Infection With Cardiovascular Disease Via Non-invasive Assessment of Endothelial Function
Brief Title: Association of Endodontic Infection With Cardiovascular Disease.
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Postgraduate Institute of Dental Sciences Rohtak (Other)
Responsible Party: Sponsor
Other Study IDs: Nishant
Record Dates: First submitted 2018-01-31; First posted 2018-02-07 (Actual); Last update posted 2018-02-07 (Actual); Status verified 2017-09

CONDITIONS: Apical Periodontitis
Keywords: Cardiovascular disease, FMD, c-IMT
MeSH Terms: conditions — Periapical Periodontitis; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Test group: Subjects having periapical disease diagnosed clinically and radiographically and free from any other systemic illness. FMD and c-IMT will be determined by ultrasound
  Interventions: Diagnostic Test: FMD and c-IMT
- Control group: Healthy subject. FMD and c-IMT will be determined by ultrasound
  Interventions: Diagnostic Test: FMD and c-IMT

INTERVENTIONS:
Diagnostic Test: FMD and c-IMT — The diameter of the target artery (right brachial artery) will be measured from two- dimensional ultrasound images, with a 70 MHz linear array transducer and a standard 128XP/10 system (Acuson, Mountain View, California, USA).
  c-IMT will be assessed by M-mode ultrasonography via a vivid 7 MHz linear array transducer and a standard 128XP/10 system (Acuson, Mountain View, California, USA) with participants in the supine position.

SUMMARY:
Chronic inflammation plays a crucial role in the genesis of atherosclerosis and at the same time promotes acute cardiovascular events. Periodontal and pulpal inflammation are two major low grade chronic inflammatory infectious disease of oral cavity. Apical periodontitis is an inflammatory process, most often chronic in nature, of endodontic origin usually occurring at or near apex of the tooth root. The scientific literature has failed to provide the potential connection between endodontic infection and CV risk. Few studies have found the possible association, yet few studies does not suggest any link. The association between chronic inflammatory lesions and endothelial dysfunction can be detected using inflammatory, invasive and non-invasive markers. Inflammatory markers such as hs-CRP and Interleukins are not cost efficient and invasive markers- Angiography and Plethysmography are unethical to use on asymptomatic subjects. Non-invasive markers such as Flow mediated dilatation (FMD) and carotid intima media thickness (c-IMT) are inexpensive, fast and safe. The rationale of our study is to check the possible association between endodontic infection and CVD using non-invasive markers.

DETAILED DESCRIPTION:
Cardiovascular Disease (CVD) is the primary non-communicable cause of global mortality killing more than 7 million people per year. Chronic inflammation plays a crucial role in the genesis of atherosclerosis which further leads to cardiovascular disease. Apical periodontitis is "an acute or chronic inflammatory lesion around the apex of a tooth caused by bacterial infection of the pulp canal system". Histologically, it is represented by a periapical inflammatory response that arises after resorption of adjacent supporting bone and local infiltration of inflammatory cells. In response to chronic inflammation, endothelium dysfunction occurs which leads to switch from a Nitric Oxide environment to a reactive oxygen dominated (ROS)-dominated inflammatory environment. The nitric oxide environment of the normal functional endothelium helps to maintain an equilibrium in the circulating system by inhibiting platelet aggregation, monocyte adhesion and vascular smooth muscle cell proliferation. Coronary endothelial dysfunction is considered an early stage of atherosclerosis and is associated with an increased risk of ischaemic cardiovascular outcomes. Several cross-sectional and longitudinal studies has shown the association of Apical periodontitis and Cardiovascular disease. Yet some studies states that there is no correlation and some showing the result is inconclusive making this link very controversial. All the studies are either hospital record based studies or they used inflammatory biomarkers for evaluating the association between endodontic infection and CVD which are very expensive.

Clinically, vasoregulation has been measured in both the coronary and peripheral circulation, using changes in vessel diameter as an index of conduit vessel endothelial function. The three most common clinically used techniques are-(a) Angiography, (b) Flow mediated dilatation (FMD), (c) and Venous plethysmography. Due to the invasive nature of angiography and plethysmography, these methods are unsuitable to be used on asymptomatic patients.

On the other hand, the non-invasive nature of the FMD allows repeated measurements over time to study the effectiveness of various interventions that may affect vascular health. The sensitivity and specificity of FMD is 95% and 37% respectively. Impaired endothelium-dependent dilatation in the coronary circulation is associated with coronary atherosclerosis and coronary risk factors and improves with risk reduction therapies. It has been shown FMD was an independent predictor of cardiovascular disease. Thus, brachial artery flow-mediated dilation prove useful to assess cardio- vascular risk, guide therapy, and judge the potential utility of new interventions for cardiovascular disease. FMD, which is most widely used non-invasive ultrasound method to assess endothelial function has been used in various interventional and cross-sectional studies depicting the link between periodontitis and endothelial dysfunction. But no such studies has been done evaluating the link between endodontic infection and endothelial dysfunction using these markers.

Another commonly used non-invasive marker these days is Carotid Intima-media thickness (IMT). c-IMT is increasingly used as a surrogate end point of vascular outcomes in clinical trials aimed at determining the success of interventions that lower risk factors for atherosclerosis and associated diseases (stroke, myocardial infarction and peripheral artery diseases). This observer dependable technique, which serves both as an early detector and a follow up tool, provides information about common carotid (CCA), bifurcation, internal (ICA) and external carotid arteries. It has been established that abnormal baseline and rapid progressive CIMT are correlated to more cardiovascular and stroke events. Every 0.1 mm increase in the CIMT was associated with a 10-15% increase in the risk of myocardial infarction, and in the same line, a 13-18 % increase in stroke events. Many interventional and cross-sectional studies have shown the link between periodontitis and c-IMT.

No prospective observational trial, to the best of our knowledge, has been done till date depicting the link between endodontic infection and cardiovascular disease using FMD and c-IMT. The aim of the present study is to depict that endodontic infection is also one of the novel risk factor of CVD using a non-invasive techniques i.e. Flow mediated dilatation (FMD) and c-IMT.

AIMS AND OBJECTIVES To depict that Endodontic infection is associated with endothelial dysfuction by measuring flow mediated dilatation (FMD) of brachial artery and carotid intima media thickness (c-IMT) of common carotid artery.

MATERIALS AND METHODS

The present study will be done in the department of Radiology, PGIMS, Rohtak and Department of Cardiology, PGIMS, Rohtak.

Study subjects will be obtained from the pool of OPD patients in the Department of Conservative dentistry and Endodontics, PGIDS, Rohtak.

METHODOLOGY 35 patients who consecutively registered for a dental checkup at the OPD and fulfilled the previously mentioned criteria will be enrolled.

Additional 35 patients who were free from clinical and radiographic evidence of AP and met the inclusion and exclusion criteria of the study will be included as contols.

All individuals aged will underwent a complete CV assessment including medical history, physical examination, blood pressure measurement and 12-lead electrocardiogram.

A complete dental examination will be performed on each patient in both groups.

DENTAL EXAMINATION A panoramic radiograph will be examined and used as initial screening . It will be followed by selected periapical radiographs taken on teeth suspected of presenting AP and in all teeth with root canal treatments or presenting extensive restorations (including prosthetic restorations) with or without previous endodontic treatment.

Periapical radiographs were taken with a radiographic unit by using a long cone paralleling technique.

By using both radiographic and intraoral evaluations the following parameters were recorded:

1. Number of teeth present
2. Number and location of restored teeth
3. Number of endodontically treated teeth
4. Number and location of teeth affected by carious processes
5. Soft tissue assessment (presence and location of swelling/sinus tracts)
6. Periodontal probing
7. Number and location of teeth with AP
8. State of the upper and lower jaws Brachial Artery Assessment Patient preparation 1) Fast at least 8-12 hours before study. 2) Should not exercise, should not ingest substances like caffeine, high fat foods, vit C or tobacco at least 4-6 hours before study.

Clinical Procedure The diameter of the target artery (right brachial artery) was measured from two- dimensional ultrasound images, with a 70 MHz linear array transducer and a standard 128XP/10 system (Acuson, Mountain View, California, USA).

Patient is placed in supine position with arm comfortably placed. Right brachial artery will be imaged above antecubital fossa in longitudinal plane.

In each study 4 scans will be taken:

Scan1 (At rest) The subject lay at rest for at least 10 min before a first resting scan will be recorded.

Then diameter of the artery will be measured from anterior to the posterior "m" line (the interface between intima media and intima adventitia)

Arterial flow velocity will be measured, by means of a pulsed doppler signal at a 70deg angle to the vessel in the centre of the artery.

Scan 2 (Endothelium dependent FMD) Increased flow was then induced by inflation of a pneumatic tourniquet to a pressure of at least 50 mm Hg above systolic pressure for 4-5 min (reactive hyperaemia).

A second scan was taken for 30 s before and 90 s after cuff deflation, including a repeat flow velocity recording for the first 15 s after cuff release.

Brachial Artery diameter will be taken 45-60 sec after cuff deflation.

Scan3 (Again at rest) At least 10 min of rest is needed after reactive hyperaemia before another image is acquired to reflect the re-established baseline conditions.

Third scan is taken at this point of time. Scan4 (Endothelium independent FMD) Then 0.4 mg of nitroglycerine (GTN) is given sublingually. (GTN will be omitted if the patient refuse or if the patient had a history of migraine headaches, systolic blood pressure <100 mm Hg, previous adverse reaction to nitrates, or critical carotid artery stenosis) After 4 min fourth and final scan will be taken. Carotid intima-media thickness (c-IMT) Common carotid artery (CCA) will be used because of its convenience and high reproducibility.

c-IMT will be assessed by M-mode ultrasonography via a vivid 7 MHz linear array transducer and a standard 128XP/10 system (Acuson, Mountain View, California, USA) with participants in the supine position.

CCA will be scanned on longitudinal two-dimensional planes. Images will be obtained at the level of distal 1.0 cm of the right CCA. When an optimal image will be obtained, it was frozen on the R wave of the electro- cardiogram and stored on videotape.

For each segment, the c-IMT of the posterior wall will be measured automatically over 200 pixels with computer-assisted electronic callipers.

Maximal right CCA thickness will be measured and used for analysis. Primary Outcome variable The primary outcome variables observed for the study will be the difference in the FMD and c-IMT of the test group and control group.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years of Male.
* Presence of apical periodontitis as assessed both clinically and radiographically (teeth with apical symptoms but without radiographic appearance of AP were not include).
* Presence of at least 25 teeth.
* Echocardiographic Left Ventricle Ejection Fraction (LVEF) value >55%.
* Hepatic and renal function within normal limits (bilirubin<1.5mg/dl; creatine<2.0mg/dl).

Exclusion Criteria:

* Presence of localized or diffuse periodontal disease.
* Presence of non-endodontic lesion in Maxilla/ mandible.
* Presence of cardiovascular risk factors(arterial hypertension, dyslipidemia, DM, obesity, smoking)
* LV hypertrophy at echocardiography previous or current CVD.
* Presence of chronic inflammatory conditions in other regions involving systemic health.
* For women, use of anticonceptive hormones.
* Systemic antibiotic treatment within the previous 3 months or any other regular medication.

Ages: 20 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Males between 20-40 years of age
Study Population: Study subjects will be obtained from the pool of OPD patients in the Department of Conservative dentistry and Endodontics, PGIDS, Rohtak.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2016-11-01 (Actual); Primary Completion 2018-03-30 (Estimated); Study Completion 2018-03-30 (Estimated)

PRIMARY OUTCOMES:
Difference in FMD and c-IMT between test and control groups. | 1 year
  The primary outcome variables observed for the study will be the difference in the FMD and c-IMT of the test group and control group.

CONTACTS AND LOCATIONS:
Locations (1):
- Post Graduate Institute of Dental Sciences, Rohtak, Haryana, India

IPD SHARING:
Plan to Share IPD: No